CLINICAL TRIAL: NCT05389397
Title: De-implementation of Outdated Colonoscopy Surveillance Interval Recommendations Among Patients With Low-risk Adenomas
Acronym: DESIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1789503-1
Record Dates: First submitted 2022-05-16; First posted 2022-05-25 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Polyp of Colon
MeSH Terms: conditions — Colonic Polyps | interventions — Community-Institutional Relations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mailed Letter (Placebo Comparator)
  Interventions: Behavioral: Outreach
- Secure Message (Active Comparator)
  Interventions: Behavioral: Outreach
- Telephone Outreach (Active Comparator)
  Interventions: Behavioral: Outreach

INTERVENTIONS:
Behavioral: Outreach — Mailed letter, secure message or telephone outreach will be used depending on arm enrolled

SUMMARY:
The purpose of this study is to compare the effectiveness of three standard of care outreach approaches (i.e., mailed letter, secure message, and telephone call) on patient adoption of the new 10-year colonoscopy surveillance interval recommendation for a random sample of health plan members who have a now-outdated 5-year surveillance interval due to a finding of 1-2 small adenomas at their prior colonoscopy. The primary study endpoint is the proportion of patients in each outreach arm who adopt the new 10-year colonoscopy surveillance interval.

ELIGIBILITY:
Inclusion Criteria:

* Kaiser Permanente Northern California (KPNC) membership>12 months
* Primary medical center is either KP San Rafael, KP San Francisco, KP San Leandro, or KP Walnut Creek
* 54-70 years of age at time of 5-year surveillance colonoscopy interval
* A baseline colonoscopy with a finding of 1-2 small tubular adenomas and are due for their 5-year surveillance procedure in 2022
* Average risk for CRC
* A valid mailing address, kp.org account (i.e., KPNC's secure messaging portal), and telephone number at time of study enrollment.

Exclusion Criteria:

* More than 12 months of membership prior to index colonoscopy, and indications that would make an individual above average risk for CRC, such as: adenoma with advanced histology on colonoscopy, adenoma >10 mm on colonoscopy, family history of CRC, prior history of colonoscopy, prior history of adenomas or colon polyp diagnoses, history of IBD, history of hereditary polyposis syndrome, 3 or more adenomas, adenoma 10 mm in size or greater, adenoma with advanced histology, and any sessile serrated polyp or traditional serrated adenoma

Ages: 54 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 604 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who respond with a 10-year surveillance interval change | 2 months following outreach intervention

SECONDARY OUTCOMES:
Percentage of patients requesting a physician appointment | 2 months following outreach intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey K Lee, MD, Study Chair — Kaiser Permanente
Locations (1):
- Kaiser Permanente San Francisco Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JK, Koripella PC, Jensen CD, Merchant SA, Fox JM, Chang SX, Dang CH, Velayos FS, Boparai ES, Evans NS, Leung LJ, Badalov JM, Quesenberry CP, Corley DA, Levin TR. Randomized Trial of Patient Outreach Approaches to De-implement Outdated Colonoscopy Surveillance Intervals. Clin Gastroenterol Hepatol. 2024 Jun;22(6):1315-1322.e7. doi: 10.1016/j.cgh.2023.12.027. Epub 2024 Jan 6. PMID 38191014